CLINICAL TRIAL: NCT04179708
Title: Effectiveness of Pain Neuroscience Education Compared to a Conventional Education for Patients With Chronic Low Back Pain : A Randomized Monocentric Trial.
Brief Title: Effectiveness of Pain Neuroscience Education Compared to a Conventional Education for Patients With Chronic Low Back Pain
Acronym: EVAL-PNE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Société Française de Physiothérapie (SFP). (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018_79; 2019-A01260-57 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2019-11-25; First posted 2019-11-27 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Chronic Low-back Pain
Keywords: Therapeutic Patient Education; Chronic Low Back Pain; Chronic Pain; Pain Neuroscience Education; Pain Neurophysiology Education; Pain biology education
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pain neuroscience education (Experimental)
  Interventions: Other: Pain Neuroscience Education; Other: Conventional education
- Conventional education (Active Comparator): patient receiving a "classical" education on spinal physiology and ergonomics
  Interventions: Other: Conventional education

INTERVENTIONS:
Other: Pain Neuroscience Education — Intervention description Patients participate in a back school program including initial and final assessment, educational activities and therapeutic activities (eg. Physiotherapy, balneotherapy, physical activity, spine ergonomics, and so on) spread over 5 days. The therapeutic activities are the same in experimental and control group, only the educational activities differ.
  The educational activities represent 4 hours of intervention, ½ hours of educative initial assessment and ½ hour of educative final assessment.
  The content of Pain Neuroscience Education (experimental group) focuses on deconstruction of patho-anatomical and biomechanical believes, and the explanation of pain from the biology. This framework allows the introduction of coping strategies (eg gradual exposure to exercise, activity and physical activity) and regulation strategy (eg fragmentation of activity, stress management, and so on).
  Arms: pain neuroscience education
Other: Conventional education — assessment, educational activities and therapeutic activities (eg. Physiotherapy, balneotherapy, physical activity, spine ergonomics, and so on) spread over 5 days. The therapeutic activities are the same in experimental and control group, only the educational activities differ.
  The educational activities represent 4 hours of intervention, ½ hour of educative initial assessment and ½ hour of educative final assessment.
  The content of conventional education (control grou) focuses on patho-anatomical and biomechanical notions. This framework allows the introduction of protection strategies (eg education on good posture, good handling techniques, physical activity and therapeutic exercise in stretch and strenghten the spine in order to protect it).

SUMMARY:
The hypothesis is that pain biology education, combined with a rehabilitation program, reduces disability to 3 months, compared to conventional spinal physiology education.

ELIGIBILITY:
Inclusion Criteria:

* Low Back Pain since more than 1 year
* Affiliated to Social Security Scheme
* Rolland Moris ≥ 8
* Start Back ≥ 4

Exclusion Criteria:

* Suspicion or proven case of serious pathology such as recent vertebral fracture (less than 6 months), infection, malignant tumors and / or radiculopathy.
* Have a history of rheumatic inflammatory disease
* Have a true radiculalgia (with or without radiculopathy)
* Have a scoliosis > 30° (if it is considered as a predominant contributor of pain's persistence).
* Rating of pain > 8/10
* Have had lumbar surgery in the past 12 months
* Have had an injection in the past 3 months
* Patients under legal protection (guardianship, curatorship)
* Pregnant patients
* Patients who are not able to understand, read or speak french
* Inability to receive informed information

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2024-02-10 (Actual); Study Completion 2024-02-10 (Actual)

PRIMARY OUTCOMES:
Functional disability level (Rolland Morris questionnaire). | At 3 months

SECONDARY OUTCOMES:
Pain rating (Numeric scale) | at baseline (pre intervention), at 5 days (post intervention), at 3 months and at 1 year
Functional disability level (Rolland Morris questionnaire) | at baseline (pre intervention), at 5 days (post intervention) and at 1 year
Functional disability level (Dallas questionnaire) | at baseline (pre intervention), at 5 days (post intervention), at 3 months and at 1 year
Negatives believes level (Fear Avoidance and Belief Questionnaire) | at baseline (pre intervention), at 5 days (post intervention), at 3 months and at 1 year
Catastrophism level (Pain Catastrophizing Questionnaire) | at baseline (pre intervention), at 5 days (post intervention), at 3 months and at 1 year
Kinesiophobia level (Tampa Scale of Kinesiophobia) | at baseline (pre intervention), at 5 days (post intervention), at 3 months and at 1 year
Anxiety and Depression level (Hospital Anxiety and Depression scale) | at baseline (pre intervention), at 5 days (post intervention), at 3 months and at 1 year
Satisfaction level (18-item of Patient Satisfaction Questionnaire) | At one year
semi-conductive interview | At 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Wieczorek, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Swynghedauw, Lille, France

REFERENCES:
- [Result] Adenis N, Wieczorek V, Corbinau S, Mortain L, Thevenon A. Pain neuroscience education is not superior to spinal physiology and ergonomics education within a short multidisciplinary rehabilitation program: A randomized controlled trial. Musculoskelet Sci Pract. 2024 Nov;74:103176. doi: 10.1016/j.msksp.2024.103176. Epub 2024 Sep 5. PMID 39260006